CLINICAL TRIAL: NCT05925985
Title: Propel Drug-Eluting Sinus Stent Family Open Cohort
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PSR Ear, Nose and Throat
Record Dates: First submitted 2023-05-19; First posted 2023-07-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Propel: Patients implanted with Propel model implants
  Interventions: Other: NA-Observational Registry
- Propel Mini: Patients implanted with Propel Mini model implants
  Interventions: Other: NA-Observational Registry
- Propel Contour: Patients implanted with Propel Contour model implants
  Interventions: Other: NA-Observational Registry

INTERVENTIONS:
Other: NA-Observational Registry — NA Observational Registry

SUMMARY:
The purpose of this study is to confirm the long-term clinical safety and performance, acceptability of identified risks, and to detect emerging risks based on factual evidence for the PROPEL family of products when used according to labeling (in patients with chronic rhinosinusitis (CRS) undergoing sinus surgery). Additionally, this study intends to collect data on use of corticosteroid-eluting implants in the European CRS population. Data collected will be used to ensure continued consistency between clinical data, the information materials supplied by the manufacturer, and the risk management documentation.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements.
* Patient has or is intended to receive or be treated with an eligible Medtronic product
* Patient is consented within the enrollment window of the therapy received, as applicable

Exclusion Criteria:

* Patient who is, or is expected to be, inaccessible for follow-up
* Participation is excluded by local law
* Patient is currently enrolled or plans to enroll in concurrent drug/device study that may confound the PSR results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European CRS population implanted with Propel implants
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Long-term safety and efficacy of corticosteroid-eluting implants in patients with CRS undergoing Functional Endoscopic Sinus Surgery (FESS) | 6 months
  The primary efficacy endpoint is Sino-Nasal Outcome Test 22 item (SNOT-22) total score change from baseline to Month 6. The SNOT-22 assesses 22 symptoms associated with Chronic Rhinosinusitis (CRS) with a value from 0 (no problem) to 5 (problem as bad as it can be). The total score is assessed by summing the score for each of the 22 items. Total SNOT-22 scores of 20 and greater in patients with CRS meet criteria defined by European Position Paper on Rhinosinusitis and Nasal Polyps 2020 (EPOS 2020) as indicated for Functional Endoscopic Sinus Surgery (FESS). Baseline SNOT-22 total scores are expected to be higher at baseline prior to FESS. A decrease in SNOT-22 score at 6 months would indicate improvement in the patient's CRS symptoms.

SECONDARY OUTCOMES:
Endoscopic evaluation | 12 months
  Endoscopic evaluation scoring from baseline to month 3, 6, and12. Endoscopic evaluation is the physician's assessment via endoscopy of the adhesion/scarring, polyps, patency, polypoid oedema, and middle turbinate lateralization of the sinuses from 0 (none) to 3-4 (most severe) prior to FESS, and following FESS and Propel stent placement at 3, 6 and 12 months. Lower scores at follow-up would indicate improvement in the patient's CRS and healing compared to baseline.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (8):
  - Saint Elisabeth Krankenhaus Köln-Hohenlind, Cologne
  - Universitätsklinikum Freiburg Klinik für Hals, Nasen und Ohrenheilkunde, Freiburg im Breisgau
  - Katholisches Krankenhaus Hagen, Hagen
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - HNO Praxis & Rhinologie Zentrum München, München
  - Universitätsklinikum Münster Klinik für Hals, Nasen und Ohrenheilkunde, Münster
  - Helios Dr Horst Schmidt Kliniken, Wiesbaden
- Imperial College Healthcare NHS Trust - Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No